CLINICAL TRIAL: NCT03854825
Title: Neutral Endopeptidase for Early Detection of Acute Kidney Injury After Cardiac Surgery
Acronym: NEPAKI-CS
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Martin Bernardi, Neutral Endopeptidase for early detection of acute kidney injury after cardiac surgery, Medical University of Vienna
Other Study IDs: 1223/2015_1.9
Record Dates: First submitted 2019-02-24; First posted 2019-02-26 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI: patients with postoperative AKI defined by KDIGO
  Interventions: Procedure: Cardiac surgery
- no AKI: patients without postoperative AKI defined by KDIGO
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery

SUMMARY:
The investigators want to investigate if the urinary biomarker neprilysin can identify cardiac surgical patients suffering from postoperative AKI within 24 hours.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common complication following cardiac surgery and significantly increases morbidity, duration of hospital stay, and mortality. The diagnosis of AKI relies on changes in serum creatinine (SCr) from a baseline value or decreases in urine output. Nevertheless changes of SCr to diagnose AKI are only reliable after a minimum of 48 hours.

Neutral endopeptidase, also called neprilysin (NEP) represents a single-pass membrane glycoprotein with zinc-dependent endopeptidase activity and a short cytosolic tail and is found in epithelia, fibroblasts, and neutrophils and in soluble form in the circulation, urine, and cerebrospinal fluid. Beside the focus of interest in cardiovascular medicine for its role in heart failure, where the inhibition of NEP by the administration of sacubitril/valsartan may achieve an improvement in patients with chronic heart failure and reduced ejection fraction, there is also thought to be a link to renal damage.

NEP is expressed in the brush border of proximal tubular cells, which is first shed in renal damage and therefore it is a marker for tubular damage when it is measurable in urine In this study the investigators want to investigate if NEP is a marker for earlier detection of AKI after elective cardiac surgery compared to the currently recommended Kidney Disease - Improved Global Outcomes (KDIGO) guidelines for acute kidney injury. Also, the investigators want to investigate at predefined time points the occurrence and the progression of tubular damage during cardio-pulmonary bypass (CPB) in a closed-meshed NEP detection.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing an elective cardiac surgical intervention

Exclusion Criteria:

* Emergency procedures
* Heart transplantation
* Elective left ventricular assist device (LVAD) implantation
* Pulmonary thrombendarterectomy
* Declined informed consent
* Age < 18 years
* Pregnant woman
* Preoperative renal replacement therapy (RRT)
* Receiving medication containing sacubitril

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective cardiac surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-10-30 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
NEP-levels | 24 hours
  Difference of NEP-levels after cardiac surgery on the first postoperative day

SECONDARY OUTCOMES:
NEP-levels | approximately 6 hours
  Difference of NEP-levels after cardiac surgery at the end of procedure
Increase of NEP | approximately 6 hours
  Time-dependent increase of NEP during CPB

CONTACTS AND LOCATIONS:
Locations (1):
- Divison of Cardiothoracic Anaesthesia and Intensive Care, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Bernardi MH, Wagner L, Ryz S, Puchinger J, Nixdorf L, Edlinger-Stanger M, Geilen J, Kainz M, Hiesmayr MJ, Lassnigg A. Urinary neprilysin for early detection of acute kidney injury after cardiac surgery: A prospective observational study. Eur J Anaesthesiol. 2021 Jan;38(1):13-21. doi: 10.1097/EJA.0000000000001321. PMID 32941200